CLINICAL TRIAL: NCT00712660
Title: ITAREPS Trial: A Prospective Randomized Double-blind Controlled Study in IT-aided Mobile Phone-based Relapse Prevention Program in Schizophrenia.
Brief Title: Study With Information Technology (IT) - Aided Preventive Program in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prague Psychiatric Center (Other Government)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Filip Spaniel, M.D., Ph.D, MD, Prague Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITA-04-2008
Record Dates: First submitted 2008-06-06; First posted 2008-07-10 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: prevention; relapse; schizophrenia
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): In the active-ITAREPS group, the e-mail ALERT message feedback to the investigator will be activated. The core study intervention was 20% antipsychotic dose increase within 24 hours in response to a Pharmacological Intervention Requiring Event (PIRE) defined as either: A) the receipt of any INITIAL ALERT (IA) e-mail. A dose increase was obligatory in such cases regardless of the current clinical status of the patient; or B) the receipt of an ALERT EMERGENCY (AE) e-mail after which the investigator confirmed clinical worsening via phone contact with the patient. AE is defined as further worsening in EWSQ scores during 3 week period after announcement of IA.
  Interventions: Drug: antipsychotic dose increase
- TAU (Placebo Comparator): In the treatment-as-usual study arm (control, non-active ITAREPS), the e-mail ALERT message feedback will not be activated. In this group, even in the presence of early warning sings, the investigators will be kept blinded to the EWSQ scores, will receive no ALERT message and thus no early pharmacologic intervention based on the ITAREPS program will be prompted. Treatment in the control group will consist of routine clinical and medication management with the frequency of visits common in the outpatient clinical settings. There will be no intevention based on ITAREPS.
  Interventions: Other: no intervention

INTERVENTIONS:
Drug: antipsychotic dose increase — 20% increase in the dose of current antipsychotic medication
  Other Names: All antipsychotics approved for clinical use in Czech and Slovak Republic:
  Arms: A
Other: no intervention — Treatment as usual
  Other Names: Treatment as usual
  Arms: TAU

SUMMARY:
Information Technology-aided Program of Relapse Prevention in Schizophrenia (ITAREPS) will decrease the number of hospitalizations in patients with schizophrenia or schizoaffective disorder who are treated in the outpatient psychiatric setting, as evidenced by the reduction of the total number of hospitalizations due to relapse of psychosis at the end of the 12-months follow-up period in the active ITAREPS group compared to the control (treatment-as-usual) group.

DETAILED DESCRIPTION:
Title of Study:

ITAREPS Trial: A Prospective Randomized Double-blind Controlled Study in IT-aided Mobile Phone-based Relapse Prevention Program in Schizophrenia.

Estimated Number of Study Centers and Countries:

30-40 outpatient psychiatrists in the Czech Republic and in the Slovak Republic.

Research Hypothesis:

Information Technology-aided Program of Relapse Prevention in Schizophrenia (ITAREPS) will decrease the number of hospitalizations in patients with schizophrenia or schizoaffective disorder who are treated in the outpatient psychiatric setting, as evidenced by the reduction of the total number of hospitalizations due to relapse of psychosis at the end of the 12-months follow-up period in the active ITAREPS group compared to the control (treatment-as-usual) group.

Study Phase:

Non Drug Interventional Study

Study Objective:

To evaluate effectiveness of the ITAREPS program in reduction of the number of hospitalizations due to relapse of psychosis. The ITAREPS program employs mobile phone communication between the psychiatrist and the patient. Subjects enrolled in the project (patient and his/her family member) are instructed to complete two separate versions of the 10-item Early Warning Signs Questionnaire (EWSQ) upon a weekly SMS request sent automatically by the system. EWSQ detects proportional worsening (or a new onset) of psychotic symptoms compared to the last week's score of the completed questionnaire. Individual EWSQ scores are sent by the subjects back to the ITAREPS system as a SMS text message. If the EWSQ score exceeds given score thresholds, an immediate ALERT requesting a therapeutic intervention is announced to the investigator as an e-mail message and a timely pharmacological intervention is triggered in accordance with the Early Intervention Algorithm (EIA).

Study design:

This is an international, randomized, double-blind, controlled, design-blinded, non drug, interventional study. Subjects (patient and family member pairs) will be randomized at a 1:1 ratio into the interventional or control group. All subjects will complete the EWSQ on a weekly basis. In the interventional group, e-mail alert message feedback to the investigator will be active and the investigator will react by using the EIA. In the control (treatment-as-usual) group, alerts will not be generated and the investigator will detect and react on the potential signs of the psychotic relapse only by using the standard clinical approach. The ALERTs will be reported to the investigators in approximately 50% of all ALERT events but the investigators and subjects will be kept blinded about the real study design - parallel or (multiple) cross-over. The type of the study design is specified only in section 3.1.1. of the protocol. This section will not be available to the investigators and will be provided only for the purpose of the regulatory and ethics review.

Study duration: 12 months

Number of subjects:

150 enrolled patient/family member pairs (i.e. 300 subjects) resulting in expected 120 evaluable patient/family member pairs (i.e. 240 subjects) will be participating in the study.

Study population:

Male and female patients between 18 to 60 having ICD-10 diagnosis of schizophrenia or schizoaffective disorder and their healthy family members, both eligible for mobile phone communicating.

Statistical Methods:

The primary effectiveness analysis will be a comparison of the upper bound of 95% confidence interval (CI) for the mean number of hospitalizations in patients in the active ITAREPS group at month 12 compared to the control (treatment-as-usual) group. Rehospitalization risk will be analyzed using Kaplan-Meier survival analysis in both groups. An interim analysis evaluating the between group differences in the number of psychiatric hospitalization days will be performed after all enrolled patients have completed their Visit 2 (month 6).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages 18 to 60 years, inclusive. Earliest inclusion day is the 18th birthday and the latest is the day before the 61st birthday.
2. A diagnosis of schizophrenia or schizoaffective disorder according to ICD-10 classification.
3. Increased risk for relapse, defined as having at least 1 psychiatric hospitalization for psychosis within the past 3 years and at least 2 psychiatric hospitalizations for psychosis in total (i.e. ≥ 2 hospitalizations).
4. Clinical Global Impression scale - Severity (CGI-S) ≤ 3 at study Visit 1.
5. All patients must be on stable doses of antipsychotic medication during the study entry.
6. Absence of organic mental disorder, mental disorder due to psychoactive substance use or mental retardation.
7. Presence of a cooperating family member, caregiver or other person who is in frequent contact with the patient (at least 4 times a week) and who is willing to participate in the trial.
8. Signed written informed consent. The informed consent process must be documented by signing the informed consent form prior to any study-related procedures.
9. Eligibility for mobile phone communicating.

Exclusion Criteria:

1. Participation in another relapse prevention program or another interventional clinical trial will be prohibited during the entire participation in the study. Subjects enrolled in observational (non-interventional) trials are not excluded from this study.
2. Hayward compliance rating scale score < 2 at Visit 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The reduction of the number of hospitalizations for psychotic relapses in patients diagnosed with schizophrenia and schizoaffective disorder | November 2008-November 2009

SECONDARY OUTCOMES:
EWSQ 10P and 10FM sensitivity, specificity, positive predictive value | November 2008-November 2009
No. of hospitalization days | November 2008-November 2009
Assessment of the natural course of the psychotic illness | November 2008-November 2009
Correlation between baseline CGI and the No. of hospitalizations at the endpoint | November 2008-November 2009

CONTACTS AND LOCATIONS:
Overall Officials: Filip Spaniel, M.D., PhD.,, Principal Investigator — Prague Psychiatrc Center
Locations (1):
- Prague Psychiatric Center, Prague, Ustavni, Czechia

REFERENCES:
- [Background] Spaniel F, Vohlidka P, Hrdlicka J, Kozeny J, Novak T, Motlova L, Cermak J, Bednarik J, Novak D, Hoschl C. ITAREPS: information technology aided relapse prevention programme in schizophrenia. Schizophr Res. 2008 Jan;98(1-3):312-7. doi: 10.1016/j.schres.2007.09.005. Epub 2007 Oct 24. PMID 17920245
- [Derived] Spaniel F, Hrdlicka J, Novak T, Kozeny J, Hoschl C, Mohr P, Motlova LB. Effectiveness of the information technology-aided program of relapse prevention in schizophrenia (ITAREPS): a randomized, controlled, double-blind study. J Psychiatr Pract. 2012 Jul;18(4):269-80. doi: 10.1097/01.pra.0000416017.45591.c1. PMID 22805901